CLINICAL TRIAL: NCT04436991
Title: Antibiotic Dosing in Geriatric Patients At the Emergency Department
Acronym: AGED
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: EC/2017/1369 (BC-01030)
Record Dates: First submitted 2020-06-09; First posted 2020-06-18 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Elderly Infection; Frailty; Frail Elderly Syndrome; Infection, Bacterial
Keywords: amoxicillin; piperacillin-tazobactam; temocillin; pharmacokinetics; pharmacodynamics
MeSH Terms: conditions — Frailty; Bacterial Infections | interventions — Blood Specimen Collection; Blood Culture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Biospecimen Retention: Samples With DNA — Whole blood, serum, plasma, blood cultures, urine samples, sputum.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Amoxicillin-clavulanate: Administration of amoxicillin-clavulanate as standard care therapy (4x or 6x 1g/d). Blood sampling in early and steady state dose (up to 5 samplings per dose). Collection of hemocultures, urine samples and sputum samples when possible.
  Interventions: Diagnostic Test: Blood sampling; Diagnostic Test: Sputum sample; Diagnostic Test: Hemoculture; Diagnostic Test: Urine sample
- Piperacillin-tazobactam: Administration of piperacillin-tazobactam as standard care therapy (4x 4g/d). Blood sampling in early and steady state dose (up to 5 samplings per dose). Collection of hemocultures, urine samples and sputum samples when possible.
  Interventions: Diagnostic Test: Blood sampling; Diagnostic Test: Sputum sample; Diagnostic Test: Hemoculture; Diagnostic Test: Urine sample
- Temocillin: Administration of temocillin as standard care therapy (2x or 3x 2g/d). Blood sampling in early and steady state dose (up to 5 samplings per dose). Collection of hemocultures, urine samples and sputum samples when possible.
  Interventions: Diagnostic Test: Blood sampling; Diagnostic Test: Sputum sample; Diagnostic Test: Hemoculture; Diagnostic Test: Urine sample

INTERVENTIONS:
Diagnostic Test: Blood sampling — At predefined time points through a venous catheter already in place. Max. volume to be withdrawn: Maximum 4ml/sample. Maximum 10 samples/patient.
  A last blood sample will be taken, if necessary, after the end of antibiotic therapy, between day 7 and day 14. Though blood results preferably will be used from available data from tests already done during standard treatment.
  Samples are collected in lithium-heparin tubes (without gel) and centrifuged immediately (within a maximum of 30 minutes after sampling) at room temperature: 8 minutes at 1885g.
  Plasma is then collected and divided in two separated labelled Eppendorf tubes 1.5 ml and immediately frozen at - 80 °C. If this is not immediately possible, tubes are frozen at - 20 °C and at regular time points transferred to a freezer at - 80 °C (minimum twice a day).
Diagnostic Test: Sputum sample — Bacteriological specimen, such as blood cultures, urine samples, sputum ea., which are usually collected in every patient according to standard care will be retained. If there is bacterial growth, MIC's will be calculated on these strains for study purpose.
Diagnostic Test: Hemoculture — Bacteriological specimen, such as blood cultures, urine samples, sputum ea., which are usually collected in every patient according to standard care will be retained. If there is bacterial growth, MIC's will be calculated on these strains for study purpose.
Diagnostic Test: Urine sample — Bacteriological specimen, such as blood cultures, urine samples, sputum ea., which are usually collected in every patient according to standard care will be retained. If there is bacterial growth, MIC's will be calculated on these strains for study purpose.

SUMMARY:
In this pilot study, we will investigate whether - with the current dosing regimens, used in the Ghent University Hospital - pharmacodynamic targets regarding beta-lactam antibiotics (more specific Amoxicilline-Clavulanate, Piperacillin-Tazobactam and Temocillin) are attained in frail patients admitted to the geriatric department.

DETAILED DESCRIPTION:
In drug research studies, older people - and especially patients with a geriatric profile or frailty risk - are very frequently excluded. Moreover, drug dosing is often extrapolated from studies in younger adults with failure to consider potential differences in pharmacokinetics (PK) and pharmacodynamics (PD).

Studies on dosing of beta-lactam antibiotics in geriatric or frail patients aged 75 years or older have, to the best of our knowledge, never been performed.

In this pilot study, we will investigate whether - with the current dosing regimens, used in the Ghent University Hospital - pharmacodynamic targets regarding beta-lactam antibiotics (more specific Amoxicilline-Clavulanate, Piperacillin-Tazobactam and Temocillin) are attained in frail patients admitted to the geriatric department.

This monocentric, prospective, observational trial is currently ongoing at the emergency department and geriatric department of the Ghent University Hospital.

Amoxicillin/clavulanic acid 1000/200mg of piperacillin-tazobactam 4000mg or temocillin 2000mg was infused intravenously over 30 minutes using a syringe pump. The standard dosing regimes were used.

An infusion catheter of minimum 18-gauge was placed in the contralateral arm to the arm in which the antibiotic dose was administered. Blood samples were collected from this catheter at first dose and assumed steady state conditions. Steady state was assumed to be reached after minimal 24h (> 4 doses at four - six hourly interval) of therapy. The goal was to obtain 5 first dose and 5 steady dose samples in every patient.

Material for bacteriological analysis, such as blood cultures, urine samples, sputum, were collected in every patient according to standard care. In case of bacterial growth, MIC's were measured on the reported strains when possible.

Amoxicillin, clavulanic acid, piperacillin, tazobactam and temocillin were measured using a validated ultra-performance liquid chromatographic method with tandem mass spectrometric detection.

Serum creatinine, cystatin C, procalcitonin, infection parameters (CRP, WBC count) and albumin were obtained from standard blood samples performed in these patients at day one and also later on during their therapy.

Three frailty score systems (KATZ, Geriatric 8 - G8, Cumulative Illness Rating Scale - CIRS) were calculated.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting at the emergency department and later on admitted to the geriatric department
* Patient age 75 years or older
* Patients with geriatric profile according to KATZ scale, G8 screening test or CIRS score.
* Patient receiving antibiotic treatment (amoxicillin-clavulanate, piperacillin-tazobactam)
* Intravenous access available for blood sampling. For measurement of the peak concentration an intravenous access other than the drug infusion line is required.

Exclusion Criteria:

* Admission to other units than the geriatric department incl. the ICU.
* Absence of informed consent
* Known hypersensitivity to beta-lactam antibiotics
* Patients who received oral amoxicillin-clavulanate prior to admission will not be included in the iv. amoxicillin-clavulanate group.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Frail elderly patients with a minimum of 75 years old, presenting at the emergency department and in need for hospitalization at the geriatric ward, in which a betalactam antibiotic treatment was started.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2018-01-03 (Actual); Primary Completion 2021-09-03 (Actual); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Blood concentrations of amoxicillin-clavulanate. | Within the first 12 hours (early dose) of treatment and after 24 - 48 hours of treatment (steady state)
  To investigate whether blood concentrations with maximum antimicrobial activity are achieved with current dosing regimens in first-dose or early-dose conditions and in steady-state conditions.
Blood concentrations of piperacillin-tazobactam. | Within the first 12 hours (early dose) of treatment and after 24 - 48 hours of treatment (steady state)
  To investigate whether blood concentrations with maximum antimicrobial activity are achieved with current dosing regimens in first-dose or early-dose conditions and in steady-state conditions.
Blood concentrations of temocillin. | Within the first 12 hours (early dose) of treatment and after 24 - 48 hours of treatment (steady state)
  To investigate whether blood concentrations with maximum antimicrobial activity are achieved with current dosing regimens in first-dose or early-dose conditions and in steady-state conditions.

SECONDARY OUTCOMES:
Measured total and unbound concentrations of beta-lactam antibiotics. | Within the first 12 hours (early dose) of treatment and after 24 - 48 hours of treatment (steady state)
  To compare measured total and unbound concentrations of beta-lactam antibiotics with predefined pharmacodynamic targets.
Response to antimicrobial therapy. | The end of individual antibiotic therapy with an average of 1 week
  To describe therapeutic response to antimicrobial therapy using procalcitonin.
Achievement of pharmacodynamic targets measured by questionnaire, vital signs, blood results and side effects. | The end of individual antibiotic therapy with an average of 1 week
  To compare achievement of pharmacodynamic targets in early-dose and steady-state conditions.
Clearance of betalactam antibiotics. | Within the first 12 hours (early dose) of treatment and after 24 - 48 hours of treatment (steady state)
  To compare clearance of betalactam antibiotics and correlate with renal function using creatinin clearance en cystatin C.

CONTACTS AND LOCATIONS:
Overall Officials: Tania Desmet, Dr., Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Students participating at the study (registered ethical committee) can consult individual participant data.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: During the whole study course.
Access Criteria: To be approved by ethical committee.